CLINICAL TRIAL: NCT01523223
Title: A Phase I Study of CD8 Memory T-Cell Donor Lymphocyte Infusion for Relapse of Hematolymphoid Malignancies Following Matched Related Donor Allogeneic Hematopoietic Cell Transplantation
Brief Title: Donor Peripheral Stem Cell Transplant in Treating Patients With Hematolymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Lowsky (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Lowsky, Associate Professor Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT243; NCI-2012-00044 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SU-01272012-9028 (Other: Stanford University); 22626 (Other: Stanford IRB)
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2016-07

CONDITIONS: Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Relapsing Chronic Myelogenous Leukemia; Splenic Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (DLI) (Experimental): Patients undergo CD8+ memory T-cell infusion over 10-20 minutes.
  Interventions: Biological: therapeutic allogeneic lymphocytes

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes — Undergo CD8 memory T-cell infusion
  Other Names: ALLOLYMPH

SUMMARY:
This phase 1 trial studies the side effects and the best dose of donor CD8+ memory T-cells in treating patients with hematolymphoid malignancies. Giving low dose of chemotherapy before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-cancer effects). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of purifying allogeneic CD8+ memory T-cells suitable for clinical application and to determine the safety and maximum tolerated dose (MTD) of these cells in patients with recurrent or refractory hematolymphoid malignancies following allogeneic hematopoietic cell transplant (HCT).

SECONDARY OBJECTIVES:

I. To determine disease response, time to disease progression, event-free survival, and overall survival following treatment with allogeneic CD8+ memory T-cells.

II. To assess donor specific chimerism before and at designated time points after treatment with allogeneic CD8+ memory T-cells.

OUTLINE: This is a dose-escalation study.

Patients undergo CD8+ memory T-cell infusion over 10 to 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have undergone a human leukocyte antigen (HLA) matched (sibling) allogeneic HCT for a hematologic or lymphoid malignancy other than chronic myelogenous leukemia (CML) who have recurrent or persistent disease and are otherwise eligible for donor leukocyte infusions CML patients with persistent disease after receiving donor lymphocyte infusion of at least 1x10^8cells/kg will be eligible for CD8+ memory T cell infusion
* Patients must have no evidence of active graft-versus-host disease and must be on a stable immunosuppressive regimen without a change in drugs dosage in the 4 weeks prior to the planned CD8+ memory T cell infusion
* Patients must not have any active infections
* Patients must have a performance status of > 70% on the Karnofsky scale
* Serum creatinine of < 2 mg/dl or creatinine clearance of > 50 cc/min
* Bilirubin of < 3 mg/dl Transaminases < 3 times the upper limit of normal
* Patients must have negative antibody serology for the human immunodeficiency virus (HIV1 and 2) and hepatitis C virus and negative test for hepatitis B surface antigen

DONOR:

* Donors must be an HLA matched sibling
* Donors must be 18-75 years of age, inclusive
* Donors must be in a state of general good health
* Donors must have a white blood cell count > 3.5 x 10^9/liter DONOR: Platelets > 150 x 10^9/liter
* Donors: Hematocrit > 35%
* Donors must be capable of undergoing leukapheresis
* Donors must not be seropositive for HIV 1 and 2, Hepatitis B surface antigen, Hepatitis B core antibody, Hepatitis C antibody, human T-lymphotropic virus (HTLV) antibody, cytomegalovirus (CMV) immunoglobulin (Ig)M, or Rapid Plasma Reagin (RPR) (Treponema)
* Female donors must not be pregnant or lactating

Exclusion Criteria:

* Diagnosis of CML except patients who have failed prior donor leukocyte infusion with a minimum cell dose of 1x10^8 cells/kg
* Patients who have been diagnosed with a second cancer (except carcinoma in situ of the cervix and basal cell carcinoma of the skin) which is currently active or has been treated within three years prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Occurrence (individual listings and summary) of dose-limiting toxicities | 60 days following CD8+ memory T-cell infusion
Incidence of GVHD | Change from Baseline to 60 days following the CD8+ memory T-cell infusion

SECONDARY OUTCOMES:
Disease response as assessed by complete remission, partial remission, stable disease, and progressive disease from radiographic and cellular or tissue samples | Change from baseline to 180 days following infusion
  Measured 90 and 180 days following infusion
Incidence of donor-specific chimerism assessed by STR analysis | Change from baseline to 6 months
  Measured monthly for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] Muffly L, Sheehan K, Armstrong R, Jensen K, Tate K, Rezvani AR, Miklos D, Arai S, Shizuru J, Johnston L, Meyer E, Weng WK, Laport GG, Negrin RS, Strober S, Lowsky R. Infusion of donor-derived CD8+ memory T cells for relapse following allogeneic hematopoietic cell transplantation. Blood Adv. 2018 Mar 27;2(6):681-690. doi: 10.1182/bloodadvances.2017012104. PMID 29572391